CLINICAL TRIAL: NCT05552781
Title: A Phase I/IIa, Open-label, Dose-escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Preliminary Anti-tumor Activity of H002 in Patients With EGFR Mutation Locally Advanced or Metastatic NSCLC
Brief Title: H002 in Patients With EGFR Mutation Locally Advanced or Metastatic NSCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RedCloud Bio (Industry)
Collaborators: R&G Pharma Studies Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H002-101CN
Record Dates: First submitted 2022-08-19; First posted 2022-09-23 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Dose-escalation and Expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- 20 mg QD, oral (Experimental): H002 20mg QD, orally administered in fasting state, receive a single dose of H002 orally, followed by a 4-day washout period. Then, the same dose of H002 will be administered QD until disease progression or not tolerated.
  Interventions: Drug: H002 capsule
- 40 mg QD, oral (Experimental): H002 40mg QD, orally administered in fasting state, receive a single dose of H002 orally, followed by a 4-day washout period. Then, the same dose of H002 will be administered QD until disease progression or not tolerated.
  Interventions: Drug: H002 capsule
- 80 mg QD, oral (Experimental): H002 80mg QD, orally administered in fasting state, receive a single dose of H002 orally, followed by a 4-day washout period. Then, the same dose of H002 will be administered QD until disease progression or not tolerated.
  Interventions: Drug: H002 capsule
- 150 mg QD, ora (Experimental): H002 150mg QD, orally administered in fasting state, receive a single dose of H002 orally, followed by a 4-day washout period. Then, the same dose of H002 will be administered QD until disease progression or not tolerated.
  Interventions: Drug: H002 capsule
- 250 mg QD, oral (Experimental): H002 250mg QD, orally administered in fasting state, receive a single dose of H002 orally, followed by a 4-day washout period. Then, the same dose of H002 will be administered QD until disease progression or not tolerated.
  Interventions: Drug: H002 capsule
- 350 mg QD, oral (Experimental): H002 350mg QD, orally administered in fasting state, receive a single dose of H002 orally, followed by a 4-day washout period. Then, the same dose of H002 will be administered QD until disease progression or not tolerated.
  Interventions: Drug: H002 capsule

INTERVENTIONS:
Drug: H002 capsule — Small molecule, Capsule
  Other Names: H002

SUMMARY:
This is a phase I/IIa, open-label, dose-escalation and expansion study to evaluate the safety, tolerability, PK and preliminary anti-tumor activity of H002 when given orally in patients with EGFR mutation-positive locally advanced or metastatic non-small cell lung cancer (NSCLC).

The study will contain two parts: Part A is dose escalation phase (i.e., Phase I) and Part B is dose expansion phase (i.e., Phase IIa).

DETAILED DESCRIPTION:
Part A (Dose Escalation Phase) Approximately 36 subjects will be enrolled, based on the "3+3" design for dose escalation and safety evaluation requirements. The total number of subjects will depend upon the number of dose escalations necessary.

Part B (Dose Expansion Phase) Up to 20 subjects will be enrolled in each expansion arm, the total number of subjects will depend upon the number of dose expansions (expansions may be at more than one dose depending upon emerging data).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 18 years at time of signing informed consent form (ICF).
2. Histological or cytological confirmed diagnosis of unresectable locally advanced or metastatic NSCLC.
3. Subjects must have NSCLC harboring one or more active EGFR mutations known to be associated with EGFR-TKI sensitivity (including, but not limited to Del19 and L858R).

   * Part A: All subjects may provide tumor sample to central laboratory to analyze the EGFR mutation status according to their own willingness;
   * Part B: All subjects must provide tumor sample to central laboratory to analyze the EGFR mutation status. And subjects must have NSCLC harboring EGFR C797S mutation.

   Note: Tumor sample can be either an archival sample or a sample obtained by pretreatment biopsy prior to H002 treatment.
4. • Part A: Subjects have received the best treatment available as determined by the physician and must have radiological documented disease progression on the last treatment administered prior to enrolling in the study.

   • Part B: Subjects have received at least one previous EGFR-TKI treatment and have radiological documented disease progression on the previous continuous EGFR-TKI treatment. In addition, subjects may have received other antitumor treatments and must have radiological documented disease progression on the last treatment administered prior to enrolling in the study.
5. Presence of at least one measurable lesion according to RECIST v1.1 per investigator assessment.
6. ECOG performance status of 0-1.
7. Life expectancy ≥ 12 weeks.
8. Adequate hematologic and organ function per protocol.
9. Women of childbearing potential (WOCBP) and fertile males with WOCBP partners must use highly effective contraception per protocol throughout the study. WOCBP must have a negative serum and/or urine pregnancy test result within 7 days prior to the first dose of H002.
10. Signed ICF, and this must be obtained before the performance of any protocol-specific procedures.

Exclusion Criteria:

1. Treatment with any of the following:

   Prior treatment with an EGFR-TKI within 8 days or approximately 5 × t1/2 prior to the first dose of H002, whichever is longer; Prior treatment with immunotherapy or biotherapy within 4 weeks prior to the first dose of H002; Radiotherapy (palliative radiotherapy is completed at least 2 weeks prior to the first dose of H002 can be enrolled) within 4 weeks prior to the first dose of H002; Herbal therapy that has anti-tumor effects within 2 weeks prior to the first dose of H002; Mitomycin and nitrosourea within 6 weeks prior to the first dose of H002; Oral fluorouracil such as tegafur and capecitabine within 2 weeks prior to the first dose of H002; Chemotherapy (except for mitomycin, nitrosourea, and fluorouracil oral drugs), or other anti-tumor drugs for the treatment of NSCLC within 4 weeks or approximately 5 × t1/2 prior to the first dose of H002, whichever is longer.
2. Subjects with EGFR exon 20 insertion mutations only.
3. Prior marketed and/or investigational treatment for EGFR C797S mutation (including, but not limited to BTP-661411, TQB3804 and BLU-945).
4. Is currently participating and receiving investigational therapy or using an investigational device, or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks or 5 × t1/2 of the investigational product, whichever is longer, prior to the first dose of H002.
5. Is expected to require any other form of anti-tumor therapy while on study.
6. Unresolved toxicity greater than CTCAE v5.0 Grade 1 from prior anti-tumor therapy.
7. ≥ CTCAE v5.0 Grade 2 skin toxicity at screening.
8. Treatment with strong inhibitors and strong inducers of CYP3A4 within 2 weeks prior to the first dose of H002, or anticipation of need for such drugs during study treatment.
9. Uncontrollable pleural effusion, ascites, or pericardial effusion.
10. Subjects who have symptomatic brain metastases, meningeal metastasis or spinal cord compression.
11. Subjects who have a chronic or active infection that required systemic treatment within 2 weeks prior to the first dose of H002.
12. Subjects who have gastrointestinal disorders that will affect oral administration or the investigator judges that the absorption of H002 will be interfered.
13. History of hypersensitivity to active or inactive excipients of H002 or drugs with a similar chemical structure or class to H002.
14. Subjects who received a diagnosis of, and/or tested positive at screening for human immunodeficiency virus (HIV).
15. Subjects with active hepatitis B.
16. Presence or history of malignancy other than NSCLC with the exception of some certain early-stage cancers.
17. Subjects who have clinically significant cardiovascular diseases that occurred within 6 months prior to the first dose of H002, include but not limited to QTc interval ≥ 450 msec (male) or ≥ 470 msec (female).
18. Major surgery or significant traumatic injury occurring within 4 weeks prior to the first dose of H002 or anticipation of need for a major surgery during the study.
19. Medical history of ILD.
20. Medical history of severe eye disease without recovery to CTCAE v5.0 Grade 0 or 1.
21. Severe gastrointestinal disease within 4 weeks prior to the first dose of H002 and did not recover to ≤ CTCAE v5.0 Grade 2.
22. Has any bleeding tendency or coagulopathy within 6 months prior to the first dose of H002.
23. Administration of a live, attenuated vaccine within 4 weeks prior to the first dose of H002 or anticipation of need for such a vaccine during the study.
24. Female subjects in pregnancy or lactation.
25. Any other circumstances that would, in the investigator's judgment, prevent the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
DOSE ESCALATION PHASE：Incidence of dose-limiting toxicities (DLTs) at Cycle 0 and Cycle1. Incidence and severity of treatment-emergent adverse events (TEAEs), with severity determined according to National Cancer Institute (NCI) CTCAE v5.0. | At the end of Cycle 1 (include 4 days in Cycle 0 and 21 days in Cycle1)
  To evaluate the safety and tolerability of H002 and to determine the maximal tolerable dose (MTD), or if possible, a dose/exposure predicted to result in optimal biological dose (OBD) or recommended phase II dose (RP2D).
DOSE EXPANSION PHASE：Objective Response Rate (ORR) | [Time Frame: Up to approximately 30 months]
  To obtain a preliminary evaluation of the anti-tumor activity at the selected dose(s) of H002 when given orally as determined according to RECIST v1.1.
DOSE EXPANSION PHASE：To evaluate the incidence and severity of TEAEs, with severity determined according to NCI CTCAE v5.0. | Up to approximately 30 months
  To evaluate the safety at the selected dose(s) of H002 when given orally.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Up to approximately 30 months
  To evaluate the pharmacokinetic (PK) characteristics of H002 when given orally following single and multiple doses.
Time to reach maximum concentration (Tmax) | Up to approximately 30 months
  To evaluate the pharmacokinetic (PK) characteristics of H002 when given orally following single and multiple doses.
Area under the plasma concentration versus time curve (AUC) | Up to approximately 30 months
  To evaluate the pharmacokinetic (PK) characteristics of H002 when given orally following single and multiple doses.
Time for half the drug concentration to be eliminated（t1/2） | Up to approximately 30 months
  To evaluate the pharmacokinetic (PK) characteristics of H002 when given orally following single and multiple doses.
DOSE ESCALATION PHASE：Objective Response Rate (ORR) | Up to approximately 30 months
  To obtain a preliminary evaluation of the anti-tumor activity of H002 when given orally as determined according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1).
Disease control rate (DCR) | Up to approximately 30 months
  To obtain a preliminary evaluation of the anti-tumor activity of H002 when given orally as determined according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1).
Duration of response (DOR) | Up to approximately 30 months
  To obtain a preliminary evaluation of the anti-tumor activity of H002 when given orally as determined according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1).
Progression-free survival (PFS) | Up to approximately 30 months
  To obtain a preliminary evaluation of the anti-tumor activity of H002 when given orally as determined according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1).
Time to progression (TTP) | Up to approximately 30 months
  To obtain a preliminary evaluation of the anti-tumor activity of H002 when given orally as determined according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1).
Overall survival (OS) | Up to approximately 30 months
  To obtain a preliminary evaluation of the anti-tumor activity of H002 when given orally as determined according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Tan, Study Director — RedCloud Bio
Locations (8):
- China (8):
  - Harbin Medical University Cancer Hospital, Haerbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Affiliated to Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No